CLINICAL TRIAL: NCT03671330
Title: Phase II Randomized, Double-blind, Placebo-controlled Study of LEE011(Ribociclib) or Placebo in Combination With Endocrine Therapy for the Treatment of Pre- and Postmenopausal Chinese Women With HR Positive, HER2-negative, Advanced Breast Cancer, Including a Subset With Pharmacokinetic Analysis.
Brief Title: Efficacy and Safety of Ribociclib in Pre- and Postmenopausal Chinese Women With HR Positive, HER2-negative, Advanced Breast Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLEE011A2206
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: HR+; HER2-; breast cancer; ribociclib; Advanced breast cancer; LEE011; pre- and postmenopausal Chinese women; HR positive; HER2-negative; Endocrine therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; Anastrozole; Letrozole; Goserelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ribociclib (Experimental): Patients in pre- and postmenopausal cohorts will be randomized in the 1:1 ratio to the experimental arm or the control arm.
  Premenopausal experimental arm: NSAI + Goserelin + Ribociclib; For pre-menopausal only, patient is an adult, female ≥ 18 years old and < 60 years old at the time of informed consent.
  It is the investigators choice for NSAI based on patient's past medical history.
  Postmenopausal experimental arm:
  Letrozole + Ribociclib
  PK Cohort: Open-label ribociclib + Letrozole treatment combination.
  For postmenopausal only, patient is an adult, female ≥ 18 years old at the time of informed consent
  Interventions: Drug: Ribociclib; Drug: NSAI: Letrozole or Anastrazole; Drug: Letrozole
- Ribociclib Placebo (Placebo Comparator): Patients in pre- and postmenopausal cohorts will be randomized in the 1:1 ratio to the experimental arm or the control arm.
  Premenopausal control arm: NSAI + Goserelin + Placebo; For pre-menopausal only, patient is an adult, female ≥ 18 years old and < 60 years old at the time of informed consent.
  It is the investigators choice for NSAI based on patient's past medical history.
  Postmenopausal control arm:
  Letrozole + Placebo For postmenopausal only, patient is an adult, female ≥ 18 years old at the time of informed consent
  Interventions: Drug: Ribociclib Placebo; Drug: Ribociclib; Drug: NSAI: Letrozole or Anastrazole; Drug: Letrozole; Drug: Goserelin

INTERVENTIONS:
Drug: Ribociclib Placebo — Film-coated tablets for oral use (200 mg x 3) form Day 1 of 21 of each 28 day cycle.
  Other Names: LEE011 Placebo
  Arms: Ribociclib Placebo
Drug: Ribociclib — Film-coated tablets for oral use (200 mg x 3) form Day 1 of 21 of each 28 day cycle.
  Other Names: LEE011
Drug: NSAI: Letrozole or Anastrazole — Letrozole: Tablets for oral use, 2.5mg daily (all days of every cycle without interruption).
  Anastrazole: Tablets for oral use, 1mg daily (all days of every cycle without interruption) For Premenopausal cohort, it is the investigators choice for NSAI based on patients past history.
  For postmenopausal and PK cohorts, all patients will be on Letrozole.
Drug: Letrozole — Letrozole: Tablets for oral use, 2.5mg daily (all days of every cycle without interruption).
Drug: Goserelin — Subcutaneous implant, 3.6mg on Day 1 of each 28 day cycle
  Arms: Ribociclib Placebo

SUMMARY:
This is a Phase II randomized, double-blind, placebo-controlled study involving premenopausal and postmenopausal Chinese women plus an open-label single arm of pharmacokinetic cohort of LEE011 in combination with Letrozole in Chinese postmenopausal women with HR+, HER2- negative advanced breast cancer.

Three cohorts of patients will be enrolled: PK cohort, premenopausal cohort, and postmenopausal cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a histologically and/or cytologically confirmed diagnosis of estrogen receptor (ER) positive and/or progesterone receptor positive breast cancer by local laboratory (based on most recently analyzed biopsy).
* Patient has HER2-negative breast cancer (based on most recently analyzed biopsy) defined as a negative in situ hybridization test or an Immunohistochemistry (IHC) status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (FISH, CISH, or SISH) test is required by local laboratory testing.
* Patient must have either:

  * Measurable disease, i.e., at least 1 measurable lesion as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria (a lesion at a previously irradiated site may only be counted as a target lesion if there is a clear sign of progression since the irradiation). OR
  * If no measurable disease is present, then at least 1 predominantly lytic bone lesion must be present (patients with no measurable disease and only 1 predominantly lytic bone lesion that has been previously irradiated are eligible if there is documented evidence of disease progression of the bone lesion after irradiation).
* Patient has ECOG performance status 0 or 1.

For premenopausal cohort:

* Patient is an adult, female ≥ 18 years old and < 60 years old at the time of informed consent and has signed informed consent before any trial related activities are conducted and according to local guidelines.
* Confirmed negative serum pregnancy test before starting study treatment or patient has had a hysterectomy.
* Patient has advanced (loco regionally recurrent not amenable to curative therapy or metastatic) breast cancer not amenable to curative therapy (e.g.

surgery and/or radiotherapy).

* Patients who received ≤ 14 days of a NSAI (letrozole or anastrozole) with or without goserelin or goserelin ≤ 28 days for advanced breast cancer prior to randomization are eligible. Patients must continue treatment with the same hormonal agent + goserelin during the study. No treatment interruption is required for these patients prior to randomization.
* Patients who have received up to 1 line of chemotherapy for advanced breast cancer and have been discontinued 28 days before randomization are eligible.

For postmenopausal cohort:

* Patient is an adult, female ≥ 18 years old at the time of informed consent and has signed informed consent before any trial related activities and according to local guidelines.
* Women with advanced (locoregionally recurrent or metastatic) breast cancer not amenable to curative therapy.

Exclusion Criteria:

* Patient who has received a prior CDK4/6 inhibitor.
* Patient with symptomatic visceral disease or any disease burden that makes the patient ineligible for endocrine therapy per the investigator's best judgment
* Patient with CNS metastases.
* Patient who has not had resolution of clinical and laboratory acute toxicities related to prior anti-cancer therapy to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 Grade ≤1.
* Patient has a known history of Human immunodeficiency Virus (HIV) infection (testing not mandatory).
* Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality
* Patient is currently receiving any of the substances as defined in the protocol that cannot be discontinued 7 days prior to the start of the treatment:

For premenopausal cohort:

* Pregnant or nursing (lactating) women.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing of study treatment and for 21 days after stopping study medication.

Note: Use of oral (estrogen and progesterone), transdermal, injected or implanted hormonal methods of contraception as well as hormonal replacement therapy is not allowed in this study.

For postmenopausal cohort:

- Patient who received any prior systemic anti-cancer therapy (including hormonal therapy and chemotherapy) for advanced breast cancer.

Note: Patients who received neo (adjuvant) therapy for breast cancer are eligible. If the prior neo (adjuvant) therapy included letrozole or anastrozole, the disease free interval must be greater than 12 months from the completion of treatment until randomization.

- Patients who received ≤ 14 days of letrozole or anastrozole for advanced disease prior to randomization are eligible.

Other protocol-defined inclusion/exclusion may apply.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 327 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Progressive free survival (PFS) based on local assessment by RECIST 1.1 guideline | The primary analysis will be conducted for pre and postmenopausal cohorts separately when approximately 100 PFS events have been observed in pre- and postmenopausal cohorts (approximately 23 months).
  Progression-free survival (PFS) is the time from date of randomization/start of treatment to the date of event defined as the first documented progression or death due to any cause. If a patient has not had an event, PFS is censored at the date of last adequate tumor assessment.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameter: Cmax | 10 months
  For PK cohort only. Maximum (peak) concentration of drug in plasma.
PK parameter: Tmax | 10 months
  For PK cohort only. Time to reach maximum plasma concentration.
PK parameter: AUC024h | 10 months
  For PK cohort only. Area under the plasma concentration curve versus time.
Overall Survival (OS) | 50 months
  For pre- and postmenopausal cohorts only. Overall Survival is defined as the time from date of randomization to date of death due to any cause.
Overall response rate (ORR) | 50 months
  For pre- and postmenopausal cohorts only. Overall response rate is defined as the proportion of patients with best overall response (BOR) of CR or PR according to RECIST 1.1
Clinical Benefit Rate (CBR) | 50 months
  For pre- and postmenopausal cohorts only. Clinical Benefit Rate is defined as percentage of patients with CR, PR per RECIST or SD lasting 24 weeks or longer, per RECIST 1.1
Time To Response (TTR) | 50 months
  For pre- and postmenopausal cohorts only. Time to response is defined as the time from the date of randomization to the first documented response either CR or PR, which must be subsequently confirmed (although date of initial response is used, not date of confirmation) according to RECIST 1.1.
Duration of Response (DoR) | 50 months
  For pre- and postmenopausal cohorts only. Duration of Response applies only to patients whose best overall response is CR or PR according to RECIST1.1.
Time to deterioration of ECOG performance status from baseline | 50 months
  For pre- and postmenopausal cohorts only. Time to definitive deterioration in ECOG performance status is defined as the time from the date of randomization to the date when ECOG performance status has definitively deteriorated by at least 1 category compared with baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- China (21):
  - Novartis Investigative Site, Hefei, Anhui
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Chongqing, Chongqing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Shengyang, Liaoning
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Kunming, Yunnan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Fuzhou
  - Novartis Investigative Site, Qingdao
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.